CLINICAL TRIAL: NCT01574339
Title: An Investigation of the Effect of Long-Term Electrical Stimulation on Lower Esophageal Sphincter (LES) Pressure and Esophageal Acid Exposure in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Effect of Long-Term Electrical Stimulation on LES Pressure and Esophageal Acid Exposure in Patients With GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoStim Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS005
Record Dates: First submitted 2012-03-22; First posted 2012-04-10 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; LES Pressure; Electrical Stimulation
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: All enrolled subjects will receive a functioning device and have stimulation delivered throughout the study.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): EndoStim LES Stimulation System
  Interventions: Device: EndoStim LES Stimulation System

INTERVENTIONS:
Device: EndoStim LES Stimulation System — The EndoStim LES Stimulation System comprises three components: an electrical stimulation lead, an implantable pulse generator (IPG) and an external programmer.
  The IPG and stimulation lead are to be implanted within the subject's body using conventional laparoscopy. The device programmer is to be used by the study investigator and/or a technical representative.

SUMMARY:
The EndoStim LES Stimulation System is an investigational device intended to improve the LES pressure and restore Lower Esophageal Sphincter (LES) function in individuals suffering from Gastroesophageal Reflux Disease (GERD).

DETAILED DESCRIPTION:
EndoStim has developed an investigational medical device specifically designed to deliver electrical stimulation to the LES and has completed two clinical feasibility studies using an external version of the EndoStim stimulation system in fifteen subjects. In these two short-term studies, electrical stimulation resulted in significant increases in LES pressure.

This study will further evaluate the safety of the procedure and its feasibility for use in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 21 - 70 years of age.
* Subject has a history of heartburn, regurgitation or both for > 12 month prompting physician recommendation of continual daily use of PPI before study entry.
* Baseline GERD HRQL heartburn score following 10-14 days off PPI which is ≥ 20 and at least 10 points higher than the on PPI score
* Subject who are on standard medical therapy for 12 months or longer and experience discomfort or who are otherwise dissatisfied with GERD symptoms
* Subjects with a GERD condition that in the opinion of the PI justifies a minimally invasive reversible procedure prior to attempting anatomical change such as Nissen fundoplication
* Subject has an American Society of Anesthesiologists (ASA) Physical Status Classification I or II (or comparable local classification if any).
* Subject has exhibited excessive lower esophageal acid exposure during 24-hour pHmetry of antisecretory therapy performed within 6 months of screening visit; pH < 4 for > 5% of total time.
* Subject has a resting LES end expiratory pressure > 5mm Hg and < 15 mm Hg on a high resolution manometry within 6 months of enrollment.
* Subject has esophagitis ≤ Grade C (LA classification) on upper endoscopy within 6 months of enrollment.
* Subject has esophageal body contraction amplitude > 30 mmHg for > 50% of swallows and > 50% peristaltic contractions on high resolution manometry.
* Subject has signed the informed consent form and is able to adhere to study visit schedule.

Exclusion Criteria:

* Subject has any non-GERD esophageal motility disorders.
* Subject has gastroparesis.
* Subject has any significant multisystem diseases.
* Subject has an autoimmune or a connective tissue disorder (e.g. scleroderma, dermatomyositis, Calcinosis-Raynaud's-Esophagus, Sclerodactyly Syndrome (CREST), Sjogren's Syndrome, Sharp's Syndrome), requiring therapy in the preceding 2 years.
* Subject has Barrett's epithelium (> M2; > C1) or any grade of dysplasia.
* Subject has a hiatal hernia larger than 3 cm.
* Subject has a body mass index (BMI) greater than 35 kg/m2.
* Subject has Type 1 diabetes mellitus
* Subject has uncontrolled Type 2 diabetes mellitus (T2DM) defined as HbA1c > 9.5 in the previous 6 months, or has T2DM for > 10 years.
* Subject has a history of suspected or confirmed esophageal or gastric cancer.
* Subject has esophageal or gastric varices.
* Subject has significant cardiac arrhythmia or ectopy or significant cardiovascular disease.
* Subject has an existing implanted electrical stimulator (e.g., pacemaker, AICD).
* Subject requires chronic anticoagulant therapy.
* Subject has dysphagia or esophageal peptic stricture, excluding Schatzki's ring.
* Subject of child-bearing potential who is pregnant or intends to become pregnant during the trial period.
* Subject is currently enrolled in other potentially confounding research.
* History of any malignancy in the last 2 years.
* History of previous esophageal or gastric surgery, including nissen fundoplication.
* Subject has any condition that, at the discretion of the investigator or sponsor, would preclude participation in the trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 24 months
  Safety will be assessed by incidence and severity of adverse events through 24 months of follow-up.

SECONDARY OUTCOMES:
Change in GERD-HRQL | Change in GERD-HRQL and RDQ questionnaire score when available from baseline (as measured off PPI) to 1, 3, 6, 12, 18 and 24 months. Heartburn and regurgitation scores will be calculated separately.
  Change from baseline in GERD-HRQL. The full title of this scale is GERD Health-Related Quality of Life (GERD-HRQL) Questionnaire. The scale is as follows, with the worst outcome scored as a 5:
  0=No Symptoms
  1. Noticeable, but not bothersome
  2. Noticeable, bothersome, but not every day
  3. Bothersome daily
  4. Bothersome and affects daily activities
  5. Incapacitating to do daily activities
Change in GERD symptoms | Changes in GERD symptoms as measured by the SF-12 questionnaire will be compared between baseline assessments and post-implant measures at 6, 12, and 24 months.
  Changes in GERD symptoms measured by the SF-12 questionnaire at 6, 12, and 24 months compared to baseline.
  The full name of the scale is SF-12v2® PRO Health Survey which is a short-form patient-reported outcome (PRO) measurement that captures physical and mental well-being across eight health domains, for a variety of diseases, conditions, and treatment groups. It's made of two main summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). the practical ranges observed in a large U.S. general population are
  * PCS: 11.1 to 69.4
  * MCS: 7.4 to 73.2 Higher scores on both PCS and MCS indicate better health
Change in GERD symptoms | Changes in GERD symptoms as measured by the patient daily symptom-diary at 3, 6, 12, 18 and 24 months Vs. baseline.
  Change from baseline GERD symptoms measured by patient diary.
Change in LES pressure | Baseline LES end expiratory pressure (LESPpre) will be compared with the end expiratory pressure (LESPpost) at 3 and 6 months.
  Change from baseline in LES baseline and expiratory pressure
Change in GI symptoms | Symptoms will be compared between baseline (as measured while on and off PPI) to 1, 3, 6, 12, 18 and 24 months.
  Change from baseline in GI symptoms (while on and off PPI)
Change in esophageal acid exposure | pH will be compared between baseline and 3, 6, 12 and 24 months.
  Change in percent 24-hour esophageal pH <4.0 at baseline compared to value at 3, 6, 12 and 24 months.
Change in esophageal acid exposure | Number of reflux events >1 minute will be compared between baseline and 3, 6, 12 and 24 months.
  Change in number of reflux events > 1 minute at baseline compared to 3, 6, 12 and 24 months.
Change in esophageal acid exposure | Number of reflux events >5 minutes will be compared between baseline and 3, 6, 12 and 24 months.
  Change in number of reflux events > 5 minutes at baseline compared to 3, 6, 12 and 24 months.
Change in medication usage | The use of antisecretory medication will be compared between baseline and 3, 6, 12, 18 and 24 months.
  Change from baseline in antisecretory medication use
Change in sleep-related quality of life | Baseline and 6, 12, and 24 months scores of Sleep quality questionnaire.
  Change from baseline in Pittsburgh Sleep Quality Index (PSQI) scores. The full name of the scale Pittsburgh Sleep Quality Index (PSQI). It is a self-report questionnaire that assesses sleep quality over a one-month time interval. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.
Change in work productivity | Baseline and 6, 12, and 24 months scores of Sleep quality and Work productivity questionnaires
  Change from baseline in Work Productivity and Activity Impairment Questionnaire scores. The Work Productivity and Activity Impairment (WPAI) Questionnaire is a 6-item instrument designed to measure impairments in work and activities over the past 7 days. It assesses four main domains:
  1. Absenteeism (work time missed)
  2. Presenteeism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivity loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity impairment It produces scores for each domain expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity

CONTACTS AND LOCATIONS:
Overall Officials: A. J. Bredenoord, Dr. med., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); T. Horbach, PD. Dr. med., Principal Investigator — Stadtkrankenhaus Schwabach, Schwabach, Germany; A. Escalona, Dr. med., Principal Investigator — Hospital Clinico de la Pontificia Universidad Catolica de Chile, Santiago, Chile; Nageshwar Reddy, M.D.,, Principal Investigator — Asian Institute of Gastroenterology
Locations (10):
- Hospital Clinico de la Pontificia Universidad Catolica de Chile, Santiago, Chile
- San Ignacio, Bogotá, Colombia
- Chinese University of Hong Kong (CUHK) / Prince of Whales, Hong Kong, Hong Kong
- Asian Institute of Gastroenterology, Hyderabad, India
- . Zalvador Zubiran National Institute of Medical Science and Nutrition, Mexico City, Mexico
- Netherlands (3):
  - AMC Amsterdam, Amsterdam
  - UMC Maastrcht, Maastricht
  - UMC Utrecht, Utrecht
- North Shore Hospital, Auckland, Takapuna, New Zealand
- St. Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sidhu AS, Triadafilopoulos G. Neuro-regulation of lower esophageal sphincter function as treatment for gastroesophageal reflux disease. World J Gastroenterol. 2008 Feb 21;14(7):985-90. doi: 10.3748/wjg.14.985. PMID 18286675
- [Background] Sanmiguel CP, Hagiike M, Mintchev MP, Cruz RD, Phillips EH, Cunneen SA, Conklin JL, Soffer EE. Effect of electrical stimulation of the LES on LES pressure in a canine model. Am J Physiol Gastrointest Liver Physiol. 2008 Aug;295(2):G389-94. doi: 10.1152/ajpgi.90201.2008. PMID 18687754
- [Derived] Kappelle WF, Bredenoord AJ, Conchillo JM, Ruurda JP, Bouvy ND, van Berge Henegouwen MI, Chiu PW, Booth M, Hani A, Reddy DN, Bogte A, Smout AJ, Wu JC, Escalona A, Valdovinos MA, Torres-Villalobos G, Siersema PD. Electrical stimulation therapy of the lower oesophageal sphincter for refractory gastro-oesophageal reflux disease - interim results of an international multicentre trial. Aliment Pharmacol Ther. 2015 Sep;42(5):614-25. doi: 10.1111/apt.13306. Epub 2015 Jul 8. PMID 26153531